CLINICAL TRIAL: NCT01937390
Title: Post-Marketing Observational Study of the Impact of Adherence to Treatment With Once-Daily Administered Long-Acting Bronchodilators (LABAs / LAMAs) on Patients Health Related Quality of Life in COPD Patients
Brief Title: Observational Study of Adherence to LABA / LAMA in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 205.517
Record Dates: First submitted 2013-09-04; First posted 2013-09-09 (Estimated); Results first posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Inhalation; Tiotropium Bromide; Hardness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- LAMA/LABA Patients
  Interventions: Drug: Tiotropium 2x2.5µg tiotropium (equivalent to 2x3.154µg tiotropium bromide monohydrate) Respimat® inhaler and cartridge Solution for inhalation; Drug: Indacterol 300 µg; Drug: Tiotropium 18µg (equivalent to 22.5µg tiotropium bromide monohydrate) HandiHaler® device Inhalation powder, hard capsule; Drug: Indacterol 150 µg

INTERVENTIONS:
Drug: Tiotropium 2x2.5µg tiotropium (equivalent to 2x3.154µg tiotropium bromide monohydrate) Respimat® inhaler and cartridge Solution for inhalation — Respimat® inhaler and cartridge Solution for inhalation
Drug: Indacterol 300 µg — inhalation powder
Drug: Tiotropium 18µg (equivalent to 22.5µg tiotropium bromide monohydrate) HandiHaler® device Inhalation powder, hard capsule — HandiHaler® device Inhalation powder, hard capsule
Drug: Indacterol 150 µg — inhalation powder

SUMMARY:
The objective of the study is to observe the effect of adherence to once-daily administered long-acting bronchodilators (long-acting ß2-agonists [LABAs] / long-acting muscarinic antagonists [LAMAs]) on patients health related quality of life (HR-QoL) and to assess the relation between symptoms improvement and adherence to Chronic Obstructive Pulmonary Disease (COPD) maintenance therapy

ELIGIBILITY:
Inclusion criteria:

1. Male or female, above 40 years of age
2. Patients clinically diagnosed of COPD with no history suggestive of asthma:

   1. by scores >=5 in the COPD Population Screener,
   2. by a clinical diagnosis of COPD made by pulmonologists or internists,
   3. by a Forced Expiratory Volume (FEV1)/ Forced Vital Capacity (FVC6) ratio of <=0.70 and a FEV1 <=80% of the predicted value as assessed by copd-6 (Vitalograph, UK);
3. Maintenance treatment-naïve COPD patients who have been prescribed once daily long-acting bronchodilators (LABAs / LAMAs) for the first time at enrolment into the study
4. Patients who are able to provide signed informed consent
5. Patients who agree to be contacted for telephone/ SMS reminders via call center

Exclusion criteria:

1. Patients with contraindications to the prescribed medication
2. Patients with any disorder that would prevent the patient from being able to complete questionnaires either verbally or by self-completion
3. Pregnant or lactating women or women of childbearing potential not using an acceptable method of contraception

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Caucasians
Sampling Method: Non-Probability Sample
Enrollment: 645 (Actual)
Dates: Start 2011-11-06 (Actual); Primary Completion 2016-10-22 (Actual); Study Completion 2016-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- CTMS MIGRATION CENTER representing all obvious CTMS Dummy Sites, Ingelheim, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 645 subjects were screened in this study, out of which 585 satisfied the selection criteria and were finally entered in to the study.
Groups:
- LAMA/LABA Patients: Patients taking once daily oral inhalation of Long-acting bronchodilators (long-acting β2-agonists [LABAs]/ long-acting muscarinic antagonists [LAMAs]) during the study period of 52 weeks.
Period: Overall Study
Arm/Group | LAMA/LABA Patients
Started | 585
Completed | 550
Not Completed | 35
Not completed — Death | 2
Not completed — Lost to Follow-up | 7
Not completed — Withdrawal by Subject | 5
Not completed — Fail to return | 21

BASELINE CHARACTERISTICS:
Population: Patients who meet all of the inclusion criteria and none of the exclusion criteria (including signing the informed consent) constituted the study population.
Arm/Group | LAMA/LABA Patients
Number analyzed (Participants) | 585
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.2 (10.1)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 115
  Male | 465
  Missing | 5

OUTCOME MEASURES:

1. Primary Outcome: Clinical COPD Questionnaire (CCQ) Total Score Change From Baseline at Month 13
Description: The Clinical COPD (Chronic Obstructive Pulmonary Disease) Questionnaire (CCQ) is a standardized, validated and reliable questionnaire (in local language) to assess the impact of treatment on health status in COPD patients. CCQ total score is calculated as the arithmetic average of 10 individual scores on a 7-point scale. CCQ total score varies from 0 (very good control) to 6 (extremely poor control). Mean change in CCQ total score from baseline at month 13 is presented along with its standard error. Change in CCQ total score is calculated for each subject as:
  CCQ total score at month 13 - CCQ total score at baseline. Baseline is defined as the first assessment after enrolment (at Month 1).
Time Frame: Baseline and 13 Month
Population: Intent-to-treat (ITT): This population set included all subjects who signed informed consent form (ICF), satisfied all inclusion and exclusion criteria and have taken at least one dose of study drug.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | LAMA/LABA Patients
Number analyzed (Participants) | 585
Units on a scale | -1.55 (0.05)

2. Primary Outcome: CCQ Total Score at Month 13 (Visit 4)
Description: Mean and standard deviation of CCQ total score is presented at month 13.
Time Frame: 13 months
Population: ITT (observed cases)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | LAMA/LABA Patients
Number analyzed (Participants) | 478
Units on a scale | 2.03 (0.95)

3. Primary Outcome: Number of COPD Exacerbations Leading to Hospitalization, Per Patient
Description: Percentage of subjects hospitalized due to COPD exacerbations exactly "n" number of times during the study period is presented. Here, "n" represents the number of times each subject is hospitalized due to COPD exacerbations.
Time Frame: 13 months
Population: ITT
Measure: Number; unit: Percentage of participants
Arm/Group | LAMA/LABA Patients
Number analyzed (Participants) | 585
Percentage of participants
  1 Exacerbation | 1.7
  2 Exacerbations | 0.7
  3 Exacerbations | 0.3
  4 Exacerbations | 0.5

4. Primary Outcome: Number of COPD Exacerbations, Per Patient
Description: Percentage of subjects experienced COPD exacerbations exactly "n" number of times during the study period is presented. Here, "n" represents the number of times each subject experienced COPD exacerbations.
Time Frame: 13 months
Population: ITT
Measure: Number; unit: Percentage of participants
Arm/Group | LAMA/LABA Patients
Number analyzed (Participants) | 585
Percentage of participants
  1 Exacerbation | 12.5
  2 Exacerbations | 3.8
  3 Exacerbations | 3.2
  4 Exacerbations | 2.2
  5 Exacerbations | 0.7
  6 Exacerbations | 0.9
  7 Exacerbations | 0.2
  9 Exacerbations | 0.2

5. Secondary Outcome: Reasons of Non-adherence to Once-daily Long-acting Bronchodilators in COPD Patients
Description: Percentage of subjects corresponding to each reason of non-adherence to once-daily long-acting bronchodilators in COPD patients are presented.
Time Frame: 13 months
Population: ITT
Measure: Number; unit: Percentage of participants
Arm/Group | LAMA/LABA Patients
Number analyzed (Participants) | 585
Percentage of participants
  Felt good and decided not to take it | 1.9
  Financial reasons | 1.2
  Felt good and forgot to take it | 0.9
  Did not experience any significant improvement | 0.2
  Ran out of medicine | 0.2
  Unable to tolerate side effects | 0.2

ADVERSE EVENTS:
Time Frame: From enrolment in the study till end of study; up to 13 months.
Description: ITT Population
Arm/Group | LAMA/LABA Patients
Serious Adverse Events (participants affected / at risk) | 10/585
Other Adverse Events (participants affected / at risk) | 0/585
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LAMA/LABA Patients (N=585)
Death (General disorders) | 5
Cardiac disorder (Cardiac disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Cerebrovascular accident (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.